CLINICAL TRIAL: NCT03740347
Title: Chronic Non-inflammatory Pains in Rheumatopediatrics
Acronym: RHUMEDOL
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180230; 2018-A02317-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-11-02; First posted 2018-11-14 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2024-10

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; chronic pain; anxiety; depression; sleepiness; quality of life
MeSH Terms: conditions — Arthritis, Juvenile; Chronic Pain; Anxiety Disorders; Depression; Sleepiness | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Juvenile idiopathic arthritis and chronic pain: Patients followed for juvenile idiopathic arthritis and chronic pain in Necker Hospital
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Response to questionnaires evaluating chronic pain and its repercussion :
  * anxiety questionnaire (Revised Children's Manifest Anxiety Scale),
  * depression questionnaire (Children's Depression Inventory score),
  * sleepiness questionnaire (Pediatric Daytime Sleepiness Scale),
  * quality of life questionnaire (Pediatric Quality of Life inventory score).
  Other Names: Evaluation of the chronic pain repercussion in juvenile idiopathic arthritis

SUMMARY:
The purpose of this study is to determine the frequency of chronic pain in adolescent with juvenile idiopathic arthritis, especially when the disease is inactive or with minimal activity.

Secondary objectives are, first to determine intensity of pain and its repercussion in daily life and second to determine risk factor of chronic pain.

DETAILED DESCRIPTION:
Juvenile idiopathic arthritis is the most frequent pathology in paediatric rheumatology clinic. Pain is an important symptom in paediatric rheumatology. It is actually poorly studied and is not evaluate in disease activity score like the Juvenile Arthritis Disease Activity Score (JADAS). It is source of handicap, social and psychological distress and greatly contribute to poor quality of life. Chronic pain is frequently multifactorial, even in inflammatory disease. In adult population, rheumatologists have shown an association between inflammatory disease like spondylarthritis or rheumatology polyarthritis and fibromyalgia.

There is no specific data on chronic pain in juvenile idiopathic arthritis. Pain is mostly evaluated by the Visual Analogue Scale (VAS) with no evaluation of pain repercussion on daily life or its chronicity. This study's primary objective is to determine the frequency of chronic pain and its relationship with disease activity. Secondaries objectives are to determine repercussion of pain in daily life, and risk factor of chronic pain.

To responded to this objective, we will conduct a transversal study in a paediatric rheumatology refence centre in Necker-Enfants malades Hospital. We will include all patients between 12 and 18 years old followed in our centre for any type of juvenile idiopathic arthritis.

Patients will be evaluated as usual by their paediatrics rheumatologist during a follow-up consultation or hospitalisation with the used of the clinical JADAS. Patient accepting to participate the study will be given a paper questionnaire evaluating chronic pain, its repercussion, anxiety (by the used of the Revised Children's Manifest Anxiety Scale (RCMAS score)), depression (by the used of the Children's Depression Inventory (CDI score)), Sleepiness (by the used of the Pediatric Daytime Sleepiness Scale (PDSS score)) and quality of life (by the used of the measurement model for the Pediatric Quality of Life inventory (PedQL score)).

ELIGIBILITY:
Inclusion Criteria:

* Child from 12 to 17 years old
* Follow-up to Necker Hospital by a rheumatologist at the reference center for juvenile idiopathic arthritis (RAISE), regardless of the form
* Not opposed to participating in the study

Exclusion Criteria:

No exclusion criteria

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients over 12 years of age followed for juvenile idiopathic arthritis in the reference center at Necker-Enfants malades Hospital (RAISE)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Frequency of chronic pain and its relationship with disease activity | Day 0
  Chronic pain will be defined by the presence of recurrent or permanent moderate pain (Visual Analogue Scale (VAS) > 3 / 10), present more than 3 days a week.
  Disease activity will be evaluated by the clinical Juvenile Arthritis Disease Activity Score (JADAS) and the definition of three groups: inactive disease, minimal disease activity and active disease.

SECONDARY OUTCOMES:
Chronic pain and disease repercussions | Day 0
  Chronic pain and disease repercussion will be assessed by a paper questionnaire evaluation repercussion on scholarship, sports, sleep and social interaction.
Repercussions of pain on patient anxiety | Day 0
  Anxiety symptoms will be assessed with the Revised Children's Manifest Anxiety Scale (RCMAS) questionnaire
Repercussions of pain on depression symptoms | Day 0
  Depression symptoms will be assessed with the Children's Depression Inventory (CDI) questionnaire
Repercussions of pain on quality of life | Day 0
  Anxiety symptoms will be assessed with the Pediatric Quality of Life inventory (PedQL) questionnaire
Repercussions of pain on patient daytime sleepiness | Day 0
  Anxiety symptoms will be assessed with the Pediatric Daytime Sleepiness Scale (PDSS score)

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Goirand, MD, PhD, Principal Investigator — AP-HP, Functional Unit of "Pain and Palliative Medicine" - Necker-Enfants malades Hospital
Locations (1):
- Functional Unit of "Pain and Palliative Medicine"- Necker-Enfants malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravelli A, Martini A. Juvenile idiopathic arthritis. Lancet. 2007 Mar 3;369(9563):767-778. doi: 10.1016/S0140-6736(07)60363-8. PMID 17336654
- [Background] Consolaro A, Ravelli A. Paediatric rheumatology: Juvenile idiopathic arthritis--are biologic agents effective for pain? Nat Rev Rheumatol. 2013 Aug;9(8):447-8. doi: 10.1038/nrrheum.2013.108. Epub 2013 Jul 2. PMID 23820859
- [Background] Tupper SM, Rosenberg AM, Pahwa P, Stinson JN. Pain intensity variability and its relationship with quality of life in youths with juvenile idiopathic arthritis. Arthritis Care Res (Hoboken). 2013 Apr;65(4):563-70. doi: 10.1002/acr.21850. PMID 22972759
- [Background] Lalloo C, Stinson JN. Assessment and treatment of pain in children and adolescents. Best Pract Res Clin Rheumatol. 2014 Apr;28(2):315-30. doi: 10.1016/j.berh.2014.05.003. PMID 24974065
- [Background] Duffield SJ, Miller N, Zhao S, Goodson NJ. Concomitant fibromyalgia complicating chronic inflammatory arthritis: a systematic review and meta-analysis. Rheumatology (Oxford). 2018 Aug 1;57(8):1453-1460. doi: 10.1093/rheumatology/key112. PMID 29788461
- [Background] McErlane F, Beresford MW, Baildam EM, Chieng SE, Davidson JE, Foster HE, Gardner-Medwin J, Lunt M, Wedderburn LR, Thomson W, Hyrich KL; Childhood Arthritis Prospective Study (CAPS). Validity of a three-variable Juvenile Arthritis Disease Activity Score in children with new-onset juvenile idiopathic arthritis. Ann Rheum Dis. 2013 Dec;72(12):1983-8. doi: 10.1136/annrheumdis-2012-202031. Epub 2012 Dec 20. PMID 23256951
- [Background] Reynolds CR. Concurrent validity of "What I think and feel:" the Revised Children's Manifest Anxiety Scale. J Consult Clin Psychol. 1980 Dec;48(6):774-5. doi: 10.1037//0022-006x.48.6.774. No abstract available. PMID 7440835
- [Background] Kovacs M. The Children's Depression, Inventory (CDI). Psychopharmacol Bull. 1985;21(4):995-8. No abstract available. PMID 4089116
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Drake C, Nickel C, Burduvali E, Roth T, Jefferson C, Pietro B. The pediatric daytime sleepiness scale (PDSS): sleep habits and school outcomes in middle-school children. Sleep. 2003 Jun 15;26(4):455-8. PMID 12841372